CLINICAL TRIAL: NCT03436667
Title: Perioperative Factors Impacting Surgical Risk and Outcomes in Children
Status: Withdrawn | Type: Observational
Why Stopped: PI left the institution
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Vidya Raman, Clinical Associate Professor, Nationwide Children's Hospital
Other Study IDs: IRB18-00068
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Surgery; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Spirometry; Reaction Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic surgery: Pediatric patients presenting for ambulatory orthopedic procedures
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Reaction Time

INTERVENTIONS:
Diagnostic Test: Spirometry — Lung volumes will be measured using spirometry.
Diagnostic Test: Reaction Time — PVT-192 Psychomotor Vigilance Task Monitor is a hand-held, self-contained system used for repetitive reaction time measurement.

SUMMARY:
This prospective study will measure various factors in children coming in for ambulatory surgery and attempt to create a scoring system that would be able to predict post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 6-18 years old having ambulatory orthopedic surgery with or without planned postoperative admission.
* Patients need to be cooperative to under spirometry testing and reaction time measurement. If unable to perform, we will assess why they were not able (non-cooperative, inability, etc)

Exclusion Criteria:

* Spinal fusion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergoing ambulatory orthopedic surgery at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Post-anesthesia care unit (PACU) length of stay | Immediately post-op
  The investigators hypothesize that spirometry performance will be associated with reduced PACU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Raman, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided